CLINICAL TRIAL: NCT01669954
Title: Prospective Study to Determine the Optimum Age for Routine DEXA Screening for Osteopenia/Osteoporosis in People With HIV Infection
Brief Title: Determination of Optimum Age for DXA Screening for Osteoporosis in HIV - The Probono 1 Study
Acronym: Probono1
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: St Thomas' Hospital, London (Other)
Responsible Party: Principal Investigator, Barry Stephen Peters, Reader and Consultant HIV Medicine, Head of Research Unit, Principle Investigator, Clinical Researcher, King's College London
Other Study IDs: RJ1 09/0329; 08/H0805/56 (Other: National Research Ethics Service)
Record Dates: First submitted 2012-08-13; First posted 2012-08-21 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Osteoporosis; Fractures; HIV Infection
Keywords: HIV; Bone mineral density; Osteoporosis; Vitamin D; Fractures
MeSH Terms: conditions — Osteoporosis; Fractures, Bone; HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Controls, females: Controls who are presumed HIV uninfected, females, aged 18 or above
- Controls, males: Controls presumed HIV uninfected, males, aged 18 or above
- HIV infected patients, males: HIV patients, males, aged 18 or above
- HIV patients,: HIV patients, females, aged 18 or above

SUMMARY:
The purpose of this study is to determine the bone mineral density in male and female patients with HIV infection according to age groups.

This will enable a practical approach to screening for osteoporosis and the management and prevention of fragility fractures in people with HIV.

In addition, all risk factors commonly associated with fragility fractures and osteoporosis are collected, as is HIV drug history.

Hence, as secondary outcomes, the associations with reduced bone mineral density can be ascertained.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or above Not pregnant Able to comply with study observations and procedures Able to give fully informed consent

Exclusion Criteria:

* Pregnant Less than 18 years of age Unable to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A randomly recruited numbers of HIV uninfected controls and HIV patients aged 18 years or above, equally matched for age, and gender.
Sampling Method: Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2009-02; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Bone mineral density at Hip | The outcome is measured within 6 months (0-6 months) after entry to the study.
  Bone mineral density as determined by DXA scanning

SECONDARY OUTCOMES:
Bone mineral density at spine (L4) | The outcome is measured within 6 months (0-6 months) after entry to the study.
  As determined by DXA scan
Any lifetime fractures reported by subjects | At any stage during persons life up to and including the last visit for the volunteer to the study.
  Self-reported fractures of any type
Vitamin D levels | The outcome is measured within 6 months (0-6 months) after entry to the study.
  Plasma vitamin D

CONTACTS AND LOCATIONS:
Overall Officials: Barry S Peters, MD PhD, Principal Investigator — King's College London
Locations (1):
- St Thomas, Hospital, London, United Kingdom